CLINICAL TRIAL: NCT02110784
Title: Proof of Concept Study of Eurartesim® in Patients With Imported Uncomplicated Plasmodium Vivax Malaria
Brief Title: Eurartesim® in Patients With Imported Uncomplicated Plasmodium Vivax Malaria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST3073-ST3074-DM13-001; 2013-003763-56 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2017-06

CONDITIONS: Malaria, Vivax
Keywords: Artemisinin based Combination Therapies; eurartesim; Dihydroartemisinin/Piperaquine
MeSH Terms: conditions — Malaria, Vivax | interventions — artenimol; piperaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eurartesim tablets (Experimental): Eurartesim 320 mg piperaquine / 40 mg dihydroartemisinin film coated tablets. one or more tablets according to the body weight, once a day dor three consecutive days.
  Interventions: Drug: Eurartesim tablets

INTERVENTIONS:
Drug: Eurartesim tablets — dosage bands: 24 to <36 kg body weight: 2 tablets a day for three consecutive days 36 to <75 kg body weight: 3 tablets a day for three consecutive days 75 to 100 kg body weight: 4 tablets a day for three consecutive days
  Other Names: dihydroartemisinin/Piperaquine

SUMMARY:
The aim of the present study is to investigate the efficacy, safety and tolerability of a therapeutic course of Eurartesim® in travellers who contracted malaria due to infection by P. vivax in endemic countries.

DETAILED DESCRIPTION:
Vivax malaria occurs throughout the tropical, subtropical and some of the temperate latitudes globally. During a primary infection some P. vivax parasites become dormant in the liver (hypnozoites) during large periods of time and might subsequently cause multiple blood-stage relapses.

The asexual stages of P. vivax are generally still sensitive to chloroquine (CQ) throughout most of the world with the exception of Indonesia and Papua New Guinea where high therapeutic failure rates ranging from 5-84% have been reported. Also, there are reports of chloroquine failure from other countries and regions where the species is endemic; in particular, the presence of CQ-resistant vivax strains is now well described in several countries, including India, Brazil, Peru and Colombia.

The treatment of the dormant stages and the prevention of relapses is reached throughout the 8-aminoquinolines (primaquine is the only commercially available in this indication).

The current treatments recommended by World Health Organization (WHO) for the radical cure of CQ-resistant vivax malaria are Artemisinin based Combination Therapies (ACTs) with partner drugs having very long half-life, combined with a two weeks regiment of primaquine (WHO, 2010).

Among a variety of suitable artemisinin-based combinations, the fixed combination of dihydroartemisinin (DHA) and piperaquine (PQP )is considered an excellent therapeutic approach since it has got all the requirements considered essential for showing a positive benefit/risk ratio in malaria therapy.

Sigma-Tau i.f.r. S.p.A. has developed a DHA+PQP formulation (Eurartesim®) manufactured according to international Good Manufacturing Practice (GMP) standards and has recently received marketing authorization in Europe via a centralized procedure by the European Medicine Agency (EMA) for uncomplicated episodes of P. falciparum malaria.

A substantial amount of data have been collected in patients with uncomplicated P. falciparum malaria treated with the DHA+PQP combination. In addition, several studies have provided evidence of high cure rate in patients with P. vivax malaria treated with DHA+PQP, however, no data are available so far on efficacy and safety of the DHA+PQP treatment in patients with imported P. vivax malaria. Acquiring data is therefore of particular importance since malaria represents an important burden among all travel-acquired illnesses considering not only the number of cases (10-20% of the imported malaria cases are due to P. vivax infection) but also the potential of a fatal outcome.

The aim of the present study is to investigate the efficacy, safety and tolerability of a therapeutic course of Eurartesim® in travellers who contracted malaria due to infection by P. vivax in endemic countries. The results of such "proof of concept" study will be used for estimating the failure rate in a precise way and to dimension one or more subsequent phase III trials of comparative efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Have read the Information for the Patient and signed the Informed Consent Form;
* Aged ≥18 years and able to swallow oral medication;
* Body weight comprised between 24 kg and 100 kg (included) for males and females;
* Uncomplicated malaria with microscopically confirmed monoinfection by Plasmodium vivax or mixed infection (i.e. infection with P. vivax and other Plasmodium species);
* Willingness to comply with the study protocol and the study visit schedule.

Exclusion Criteria:

* Participation in any investigational drug study during the previous 30 days;
* Antimalarial treatment with chloroquine and quinine within the previous 6 weeks, with piperaquine-based compounds or mefloquine or lumefantrine within the previous 3 months and with halofantrine within the previous 30 days prior to screening;
* P. vivax/Plasmodium species asexual stage parasitaemia ≥ 5% Red Blood Cells (in cases of mixed infection);
* Clinical and/or laboratory features of severe malaria according to WHO criteria (WHO 2010);
* ECG abnormality that requires urgent management (i.e. clinically significant arrhythmias, Atrio-Ventricular block II and III degree etc.);
* Family history of sudden death, or known congenital prolongation of the QT interval
* Lengthening of QT interval on ECG: corrected QT interval (Fridericia's correction) ≥450 ms for males and ≥470 ms for females;
* Concomitant administration of any treatment which can induce a lengthening of QT interval (i.e. antihistamines, macrolides, etc.) and of any antimalarial drugs (for the full list of prohibited drugs refer to section 8.3);
* Any contraindication to blood sampling (i.e. important haemorrhagic diathesis);;
* Presence of intercurrent illness or any condition (i.e. severe vomiting and dehydration) which in the judgement of the Investigator would place the patient at undue risk or interfere with the study results;
* Hypoglycaemia (blood glucose levels < 2.2 mmol/L or < 40 mg/dL);
* Splenectomy;
* Pregnant or lactating women. During the study period (Day 0- Day 42), fertile women who are sexually active must use an adequate birth control method. They should utilize oral or patch contraceptives, contraceptive implant or depot injection or an intrauterine device from at least one month before screening and during the whole study period. In all the other cases they have to agree to remain inactive or use condoms with a spermicidal agent during the study period;
* Presence of jaundice;
* Known renal impairment (serum creatinine > 2X the upper limit of the hospital laboratory reference range);
* Known liver insufficiency (AST and/or ALT > 3X the upper limit of the hospital laboratory reference range);
* Relevant anaemia (Hb< 8 g/dL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-06-18 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Uncorrected adequate clinical and parasitological response (ACPR) | 21 days after the start of treatment
  The uncorrected ACPR will be considered met for all those patients that are not presenting parasitaemia and fever at day 21 follow-up visit.

SECONDARY OUTCOMES:
Proportion of aparasitaemic patients | at day 1, 2, 3, 7, 21, 42
  to evaluate efficacy of the treatment to clear blood from parasites
Proportion of afebrile patients | at day 1, 2, 3, 7, 21, 42
  to evaluate the efficacy of eurartesim in reducing fever caused by malaria
uncorrected ACPR | at day 42
Number of Patients with Serious and Non-Serious Adverse Events | up to 42 days from starting of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hatz, Prof Dr Med, Study Chair — Medical and Diagnostic Service Department, Swiss Tropical and Public Health Institute, Basel - Switzerland
Locations (13):
- Hôpital St André-CHU, Médecine interne et Maladies tropicales, Bordeaux, France
- Germany (2):
  - Medizinische Klinik mit Schwerpunkt Infektiologie, Charite/Campus Virchow-Klinikum, Berlin
  - Department of Infectious Diseases & Tropical Medicine, University of Munich, Munich
- 15. The Center for Geographic Medicine and Tropical Diseases, Department of Medicine C - The Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (4):
  - Clinica di Malattie Infettive e Tropicali, Universitá di Brescia, Brescia
  - Azienda ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliera Arcispedale S. Maria Nuova IRCCS - Dip. Medicina Interna e Spec. Mediche, Reggio Emilia
  - Centro di Malattie Tropicali - INMI Spallanzani, Roma
- Dep. Infectious Disease, Section Travel Medicine, Leiden University Medical Centre, Leiden, Netherlands
- Spain (2):
  - CRESIB-Hospital Clinic, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
- Switzerland (2):
  - Medical and Diagnostic Service Department, Swiss Tropical and Public Health Institute, Basel
  - Bern University Hospital, Bern

REFERENCES:
- [Background] Hasugian AR, Purba HL, Kenangalem E, Wuwung RM, Ebsworth EP, Maristela R, Penttinen PM, Laihad F, Anstey NM, Tjitra E, Price RN. Dihydroartemisinin-piperaquine versus artesunate-amodiaquine: superior efficacy and posttreatment prophylaxis against multidrug-resistant Plasmodium falciparum and Plasmodium vivax malaria. Clin Infect Dis. 2007 Apr 15;44(8):1067-74. doi: 10.1086/512677. Epub 2007 Mar 5. PMID 17366451
- [Background] Ratcliff A, Siswantoro H, Kenangalem E, Maristela R, Wuwung RM, Laihad F, Ebsworth EP, Anstey NM, Tjitra E, Price RN. Two fixed-dose artemisinin combinations for drug-resistant falciparum and vivax malaria in Papua, Indonesia: an open-label randomised comparison. Lancet. 2007 Mar 3;369(9563):757-765. doi: 10.1016/S0140-6736(07)60160-3. PMID 17336652
- [Background] Sinclair D, Gogtay N, Brand F, Olliaro P. Artemisinin-based combination therapy for treating uncomplicated Plasmodium vivax malaria. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD008492. doi: 10.1002/14651858.CD008492.pub2. PMID 21735431